CLINICAL TRIAL: NCT04574661
Title: Comparison of Intermittent Occlusion and Static Stretching of Muscles in Prevention of Soreness and Vital Changes in Young Adults
Brief Title: Comparison of Intermittent Occlusion and Static Stretching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC/00240 Urooj Fatima
Record Dates: First submitted 2020-09-16; First posted 2020-10-05 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Muscle Soreness
Keywords: Muscle soreness; Vital Signs; Intermittent occlusion; Static stretching
MeSH Terms: conditions — Myalgia | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static stretching (Active Comparator): Static stretching to lower limb muscles
  Interventions: Other: Static Stretching
- Intermittent occlusion (Experimental): Intermittent occlusion to lower limb
  Interventions: Other: Intermittent Occlusion

INTERVENTIONS:
Other: Static Stretching — In Control group all the individuals will be asked to perform static stretching for 10 mints, 1 set . Vitals will be monitored from every individual. On 3rd day to this protocol leg circumference, ROM of planter and dorsal flexion and numeric pain rating scale (NPRS ) will be measured alone with all the Vitals from every individual.
  Arms: Static stretching
Other: Intermittent Occlusion — Individuals of Interventional group will be asked to lay down in supine position, apply proximal thigh cuff, 220mg for 12 minutes for intermittent occlusion. During this procedure discomfort will be checked on numeric pain rating scale, if we get 6 on scale, will stop the occlusion. Vitals will be monitored from every individual. On 3rd day to this protocol leg circumference, ROM of planter and dorsal flexion and numeric pain rating scale (NPRS ) will be measured alone with all the Vitals from every individual
  Arms: Intermittent occlusion

SUMMARY:
To determine changes in Vitals caused by Intermittent Occlusion ( 220 mg ) and to compare the effectiveness of Intermittent Occlusion and Static Stretching of the lower limb muscle group in preventing the development of exercise induce Muscle Soreness

DETAILED DESCRIPTION:
Main purpose of this study is to determine changes in Vitals caused by Intermittent Occlusion ( 220 mg ) and to compare the effectiveness of Intermittent Occlusion and Static Stretching of the lower limb muscle group in preventing the development of exercise induce Muscle Soreness. As muscle soreness is very major and basis problem of every individual , specially after enrolling into some physical activity .

First consent form will be given to both male and female participants from 18 to 25 years of age and after that PAR-Q Questionnaire will be filled for every individual, so that we will check their readiness for the Exercise then all the four Vitals will measured from every individual .They will randomly assigned by lottery method to intervention group and control group. Both group individuals will be exerted by Warm up for 5 mints, heel raise in 3 sets for 10 to 15 mints until we get 4 on RPE scale, by asking to hold dumbbells of 2 kg on both of the hands. Rate of perceived exertion (RPE) is calculated by Borg grading scale .Plus, leg circumference, ROM of planter and dorsal flexion and numeric pain rating scale (NPRS) will be measured for comparison within and between the groups. Again vitals will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age limit: 18 -25 years of age.
* Both Males and Females.
* Participants intending to join a fitness or body building program shortly ( the first exercise session would be utilized to induce mild muscle soreness )
* Participants ready for physical exertion according to PAR-Q.

Exclusion Criteria:

* Obesity (body mass index ≥ 30 kg/m2).
* Skeletal or Orthopedic Injuries.
* Known Cardiovascular disease.
* Open wounds.
* Uncontrolled Hypertension (resting brachial blood pressure ≥ 140/90 mmHg).
* Exercise induced muscle soreness in last 6 months.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | 4th day
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain). It has been shown that a composite scoring system including best, worse, and current level of pain. 27 Recent studies showed that the Majority of patients of all ages and both genders prefer NRS 28. Patients feel this scale of pain measuring technique quite easy and understandable. The benefit of the NRS is that it is validated as well as quick and easy to use.
Goniometer | 4th day
  A goniometer is an instrument which measures the available range of motion at a joint. This can be an indicator of stress which is unavoidable. Many studies showed that The universal goniometer are reliable in repeated measures of joint angles 30 .Manual goniometers can be used with confidence for longitudinal assessments in the clinic
Measuring Tape | 4th day
  Tape measurement has been used for decades round measurement or the contour of the Muscle to detect atrophy or hypertrophy of Joint to determine swelling. Research shows that measuring tape is valid and reliable tool for circumference measurements .Circumference measurements taken by spring tape have high reliability
Borg Rate of Perceived Exertion | 4th day
  Research suggest that the Borg CR-10 scale is valid and reliable for monitoring exercise intensity
PAR-Q Questionnaire | 4th day
  Physical Activity Readiness Questionnaire (PARQ) clearance has been recommended prior to low-to-moderate exercise involvement. Physical Activity Readiness Questionnaire (PARQ) is safe and effective means of risk stratification for patients interested in becoming more physically active. These results support the concurrent validity of the PARQ and suggest the revisions have had their intended effect
Temperature | 4th day
  A valid Tool for temperature measurement which has been in use from centuries is Mercury Thermometer.
Pulse rate | 4th day
  The pulse rate is a measurement of the heart rate, or the number of times the heart beats per minute which can be felt by the beats by firmly pressing on the arteries, which are located close to the surface of the skin at certain points of the body. In this study we will be using Radial Artery.
Respiratory Rate | 4th day
  The respiration rate is the number of breaths a person takes per minute , when a person is at rest counting the number of breaths for one minute by counting how many times the chest rises.
Blood pressure | 4th day
  The aneroid monitor is valid and cost effective tool which for measuring blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Anam Aftab, Phd*, Principal Investigator — Riphah college of rehabilitation and allied health sciences - Rawalpindi
Locations (1):
- Shalimar Club, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magoffin RD, Parcell AC, Hyldahl RD, Fellingham GW, Hopkins JT, Feland JB. Whole-Body Vibration as a Warm-up Before Exercise-Induced Muscle Damage on Symptoms of Delayed-Onset Muscle Soreness in Trained Subjects. J Strength Cond Res. 2020 Apr;34(4):1123-1132. doi: 10.1519/JSC.0000000000002896. PMID 30399118
- [Background] Brandner CR, Warmington SA. Delayed Onset Muscle Soreness and Perceived Exertion After Blood Flow Restriction Exercise. J Strength Cond Res. 2017 Nov;31(11):3101-3108. doi: 10.1519/JSC.0000000000001779. PMID 28118308
- [Background] Hedayatpour N, Arendt-Nielsen L, Falla D. Facilitation of quadriceps activation is impaired following eccentric exercise. Scand J Med Sci Sports. 2014 Apr;24(2):355-62. doi: 10.1111/j.1600-0838.2012.01512.x. Epub 2012 Aug 12. PMID 22882137
- [Background] Kanda K, Sugama K, Hayashida H, Sakuma J, Kawakami Y, Miura S, Yoshioka H, Mori Y, Suzuki K. Eccentric exercise-induced delayed-onset muscle soreness and changes in markers of muscle damage and inflammation. Exerc Immunol Rev. 2013;19:72-85. PMID 23977721
- [Background] Dupuy O, Douzi W, Theurot D, Bosquet L, Dugue B. An Evidence-Based Approach for Choosing Post-exercise Recovery Techniques to Reduce Markers of Muscle Damage, Soreness, Fatigue, and Inflammation: A Systematic Review With Meta-Analysis. Front Physiol. 2018 Apr 26;9:403. doi: 10.3389/fphys.2018.00403. eCollection 2018. PMID 29755363
- [Background] Newton MJ, Morgan GT, Sacco P, Chapman DW, Nosaka K. Comparison of responses to strenuous eccentric exercise of the elbow flexors between resistance-trained and untrained men. J Strength Cond Res. 2008 Mar;22(2):597-607. doi: 10.1519/JSC.0b013e3181660003. PMID 18550979
- [Background] Graven-Nielsen T, Arendt-Nielsen L. Induction and assessment of muscle pain, referred pain, and muscular hyperalgesia. Curr Pain Headache Rep. 2003 Dec;7(6):443-51. doi: 10.1007/s11916-003-0060-y. PMID 14604503
- [Background] Chapman D, Newton M, Sacco P, Nosaka K. Greater muscle damage induced by fast versus slow velocity eccentric exercise. Int J Sports Med. 2006 Aug;27(8):591-8. doi: 10.1055/s-2005-865920. PMID 16874584
- [Background] Costello JT, Baker PR, Minett GM, Bieuzen F, Stewart IB, Bleakley C. Whole-body cryotherapy (extreme cold air exposure) for preventing and treating muscle soreness after exercise in adults. Cochrane Database Syst Rev. 2015 Sep 18;2015(9):CD010789. doi: 10.1002/14651858.CD010789.pub2. PMID 26383887
- [Background] Luetmer MT, Do A, Canzanello NC, Bauer BA, Laskowski ER. The Feasibility and Effects of Acupuncture on Muscle Soreness and Sense of Well-being in an Adolescent Football Population. Am J Phys Med Rehabil. 2019 Nov;98(11):964-970. doi: 10.1097/PHM.0000000000001226. PMID 31135462
- [Background] Farias Junior LF, Browne RAV, Frazao DT, Dantas TCB, Silva PHM, Freitas RPA, Aoki MS, Costa EC. Effect of Low-Volume High-Intensity Interval Exercise and Continuous Exercise on Delayed-Onset Muscle Soreness in Untrained Healthy Males. J Strength Cond Res. 2019 Mar;33(3):774-782. doi: 10.1519/JSC.0000000000002059. PMID 28614163
- [Background] Beaven CM, Cook CJ, Kilduff L, Drawer S, Gill N. Intermittent lower-limb occlusion enhances recovery after strenuous exercise. Appl Physiol Nutr Metab. 2012 Dec;37(6):1132-9. doi: 10.1139/h2012-101. Epub 2012 Sep 12. PMID 22970789
- [Background] Page W, Swan R, Patterson SD. The effect of intermittent lower limb occlusion on recovery following exercise-induced muscle damage: A randomized controlled trial. J Sci Med Sport. 2017 Aug;20(8):729-733. doi: 10.1016/j.jsams.2016.11.015. Epub 2017 Jan 24. PMID 28153608
- [Background] LaRoche DP, Connolly DA. Effects of stretching on passive muscle tension and response to eccentric exercise. Am J Sports Med. 2006 Jun;34(6):1000-7. doi: 10.1177/0363546505284238. Epub 2006 Feb 13. PMID 16476913
- [Background] Cheung K, Hume P, Maxwell L. Delayed onset muscle soreness : treatment strategies and performance factors. Sports Med. 2003;33(2):145-64. doi: 10.2165/00007256-200333020-00005. PMID 12617692
- [Background] Xie Y, Feng B, Chen K, Andersen LL, Page P, Wang Y. The Efficacy of Dynamic Contract-Relax Stretching on Delayed-Onset Muscle Soreness Among Healthy Individuals: A Randomized Clinical Trial. Clin J Sport Med. 2018 Jan;28(1):28-36. doi: 10.1097/JSM.0000000000000442. PMID 28742609